CLINICAL TRIAL: NCT03523169
Title: The Correlation of Regional Cerebral Oxygen Saturation(rScO2) Variation in Passive Leg Raising (PLR) With Neurological Outcomes of Sepsis and Septic Shock Patients
Brief Title: Cerebral Oxygen Challenge of Passive Leg Raising Test in Sepsis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-1475
Record Dates: First submitted 2018-04-11; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness; Sepsis; Cerebral Injury
Keywords: Septic associated encephalopathy; Cerebral oxygenation; Prognosis; Passive leg raising
MeSH Terms: conditions — Critical Illness; Sepsis; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis related cerebral dysfunction was underestimated in critical illness setting, and inflammatory response of brain could not be monitored directly and cerebral oximetry offered information of cerebral dysfunction. We had hypothesized cerebral oxygenation responsiveness during passive leg raising could in some way had association in predicting with the outcomes of septic shock.

DETAILED DESCRIPTION:
Research question: Does increased regional cerebral oxygen saturation variation in passive leg raising(PLR) associated with better neurological outcomes of sepsis and septic shock patients?

Specific aims:

1. To stablish an algorithm to assess focal neurological dysfunction through regional cerebral oxygen saturation(rScO2) of sepsis and septic shock patients
2. To assess the safety and gain some experiences evaluate cerebral oxygen in passive leg raising and fluid expansion.
3. To test the correlation of rScO2 variation with neurological complication and prognosis of septic shock patients.

Significance:

1. Sepsis and septic shock were associated with increased risk of mortality, elevated morbidity rates, and neuro-developmental disability.
2. The definition of SEPSIS 3.0, signify qSOFA scores as a bedside prompt that may identify patients with suspected infection who are at greater risk for a poor outcome, It uses three criteria, including altered mentation (Glasgow coma scale<15).
3. Previously, sepsis related cerebral dysfunction was underestimated in critical illness setting, and inflammatory response of brain, such as oxygen deficit of brain tissue could not be monitored directly, thus cerebral oximetry monitoring could be used for the evaluation of cerebral tissue oxygenation in real time, providing indirect information of the brain function during sepsis and septic shock.
4. Length of reduced cerebral oxygen saturation was confirmed associated with worse outcome after major surgery perioperatively. We hypothesized that cerebral oxygen metabolism was degenerated during sepsis and septic shock, and lower cerebral oxygenation would have somewhat correlations with worse outcome of sepsis and septic shock patients.

Study Design： This will be a observational cohort trial. The schematic diagram of the study is as Figure 1. Subjects will be enrolled, and then be followed up. The outcome variables will be recorded. Inclusion criteria were age above 18 either under 80 years, and diagnosed with sepsis, using Sepsis 3.0 criteria.

Whereas exclusion criteria were patients who were under 18 or above 80 years, pregnant, brain dead, severe head trauma, patients who had a difference more than 10% between the 2 probes of cerebral oxygen saturation monitor due to possible unilateral focal pathology, and whose cousins made decision to withdraw from resuscitation.

The baseline parameters of sepsis and septic shock patients are collected: demographic data (age, sex, comorbidities, resources and diagnosis), Acute Physiology and Chronic Health Evaluation (APACHE) II score (on admission and after 24 hours), hemo-dynamic parameters (mean arterial pressure [MAP], heart rate, cardiac index [CI], stroke volume variation, and global end-diastolic index using PICCO Monitor from Pulsion, Germany), serial lactic acid measurements at presentation and after 48 hours, blood gases (arterial and central venous [at presentation and every 8 hours]), and rScO2 (at presentation and every 8 hours). Delirium were diagnosed using CAM-ICU criteria for delirium in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 either under 80 years, and diagnosed with sepsis, using Sepsis 3.0 criteria.

Exclusion Criteria:

* Patients who were under 18 or above 80 years, pregnant, brain dead, severe head trauma, patients who had a difference more than 10% between the 2 probes of cerebral oxygen saturation monitor due to possible unilateral focal pathology, and whose cousins made decision to withdraw from resuscitation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The baseline parameters of sepsis and septic shock patients are collected
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Deilirium | 7 days
  Delirium, also known as acute confusional state, is an organically caused decline from a previously baseline level of mental function.It typically involves other cognitive deficits, changes in arousal (hyperactive, hypoactive, or mixed), perceptual deficits, altered sleep-wake cycle, and psychotic features such as hallucinations and delusions. Our every patient gets checked for delirium every day (usually twice or more a day) using a validated clinical tool of Confusion Assessment Method for the ICU (CAM-ICU).The first step to assessing consciousness is to assess level of consciousness.The next step is assessment of content of consciousness. Think: rapid onset, inattention, clouded consciousness (bewildered), fluctuating.

SECONDARY OUTCOMES:
28-day survival | 28 days
  28-day survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoting Wang, MD, Study Director — Peking Unioin Medical College Hospital Critical Care Medicine Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pierrakos C, Attou R, Decorte L, Velissaris D, Cudia A, Gottignies P, Devriendt J, Tsolaki M, De Bels D. Cerebral perfusion alterations and cognitive decline in critically ill sepsis survivors. Acta Clin Belg. 2017 Feb;72(1):39-44. doi: 10.1080/17843286.2016.1191851. Epub 2016 Jun 3. PMID 27352195
- [Result] Cherpanath TG, Hirsch A, Geerts BF, Lagrand WK, Leeflang MM, Schultz MJ, Groeneveld AB. Predicting Fluid Responsiveness by Passive Leg Raising: A Systematic Review and Meta-Analysis of 23 Clinical Trials. Crit Care Med. 2016 May;44(5):981-91. doi: 10.1097/CCM.0000000000001556. PMID 26741579
- [Result] Elting JW, Aries MJ, van der Hoeven JH, Vroomen PC, Maurits NM. Reproducibility and variability of dynamic cerebral autoregulation during passive cyclic leg raising. Med Eng Phys. 2014 May;36(5):585-91. doi: 10.1016/j.medengphy.2013.09.012. Epub 2013 Oct 29. PMID 24176834
- [Result] Pfister D, Siegemund M, Dell-Kuster S, Smielewski P, Ruegg S, Strebel SP, Marsch SC, Pargger H, Steiner LA. Cerebral perfusion in sepsis-associated delirium. Crit Care. 2008;12(3):R63. doi: 10.1186/cc6891. Epub 2008 May 5. PMID 18457586
- [Result] Schramm P, Klein KU, Falkenberg L, Berres M, Closhen D, Werhahn KJ, David M, Werner C, Engelhard K. Impaired cerebrovascular autoregulation in patients with severe sepsis and sepsis-associated delirium. Crit Care. 2012 Oct 4;16(5):R181. doi: 10.1186/cc11665. PMID 23036135
- [Result] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Result] Wood M, Song A, Maslove D, Ferri C, Howes D, Muscedere J, Boyd JG. Brain Tissue Oxygenation in Patients with Septic Shock: a Feasibility Study. Can J Neurol Sci. 2016 Jan;43(1):65-73. doi: 10.1017/cjn.2015.280. Epub 2015 Sep 4. PMID 26338150
- [Result] Steppan J, Hogue CW Jr. Cerebral and tissue oximetry. Best Pract Res Clin Anaesthesiol. 2014 Dec;28(4):429-39. doi: 10.1016/j.bpa.2014.09.002. Epub 2014 Sep 28. PMID 25480772
- [Result] Harilall Y, Adam JK, Biccard BM, Reddi A. The effect of optimising cerebral tissue oxygen saturation on markers of neurological injury during coronary artery bypass graft surgery. Heart Lung Circ. 2014 Jan;23(1):68-74. doi: 10.1016/j.hlc.2013.07.002. Epub 2013 Jul 30. PMID 23911209
- [Result] Maldonado Y, Singh S, Taylor MA. Cerebral near-infrared spectroscopy in perioperative management of left ventricular assist device and extracorporeal membrane oxygenation patients. Curr Opin Anaesthesiol. 2014 Feb;27(1):81-8. doi: 10.1097/ACO.0000000000000035. PMID 24366053
- [Result] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364
- [Result] Fischer GW, Lin HM, Krol M, Galati MF, Di Luozzo G, Griepp RB, Reich DL. Noninvasive cerebral oxygenation may predict outcome in patients undergoing aortic arch surgery. J Thorac Cardiovasc Surg. 2011 Mar;141(3):815-21. doi: 10.1016/j.jtcvs.2010.05.017. Epub 2010 Jun 25. PMID 20579669
- [Result] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242